CLINICAL TRIAL: NCT05406206
Title: A Phase II Study of Hepatic Arterial Infusion Chemotherapy (HAIC) Combined With Fruquintinib as Third-line Therapy for Patients With Unresectable Colorectal Cancer Liver Metastases
Brief Title: Hepatic Arterial Infusion Chemotherapy With Fruquintinib for Colorectal Cancer Liver Metastases As Third-line Therapy
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking University Cancer Hospital & Institute (Other)
Responsible Party: Principal Investigator, Zhu Xu, Chief physician, Peking University Cancer Hospital & Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Fru-HAIC-01
Record Dates: First submitted 2022-06-01; First posted 2022-06-06 (Actual); Last update posted 2022-06-06 (Actual); Status verified 2022-06

CONDITIONS: Advanced Colorectal Carcinoma; Liver Metastasis Colon Cancer
Keywords: Hepatic Arterial Infusion Chemotherapy; HAIC; Fruquintinib
MeSH Terms: interventions — HMPL-013

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HAIC combined with Fruquintinib (Experimental): HAIC with fruquintinib until progression. Fruquintinib should be administrated within 1 week after HAIC.
  Interventions: Drug: Fruquintinib; Procedure: Hepatic Arterial Infusion Chemotherapy

INTERVENTIONS:
Drug: Fruquintinib — Fruquintinib is a capsule in the form of 1mg and 5mg, once a day, 3 week on/1 week off.
  Other Names: HMPL-013
Procedure: Hepatic Arterial Infusion Chemotherapy — HAIC is a locoregional therapy for colorectal cancer liver metastasis. Oxaliplatin 85 mg/m*2 + 5-FU 2000 mg/m*2, Q4W
  Other Names: HAIC

SUMMARY:
Fruquintinib (HMPL-013) is a novel oral small molecule that selectively inhibits vascular endothelial growth factor receptors (VEGFR) 1, 2, and 3 and has demonstrated potent inhibitory effects on multiple human tumor xenografts. Combined with hepatic arterial infusion chemotherapy (HAIC), this study is conducted to assess the efficacy and safety of this regimen in patients with unresectable colorectal cancer liver metastases as the third-line therapy.

DETAILED DESCRIPTION:
This will be a single-arm, open-label, phase II study. This study will be divided into 2 stages: dose exploration and dose expansion. In the dose exploration stage, "3+3 dose escalation" design will be applied to determined the maximum tolerated dose (MTD) of fruquintinib for next stage:

Cohort A: HAIC + fruquintinib 3mg QD, 3 weeks on/1 week off (3w/1w). Cohort B: HAIC + fruquintinib 4mg QD, 3w/1w. Cohort C: HAIC + fruquintinib 5mg QD, 3w/1w.

All subjects of this study will be permitted to continue therapy with only safety monitoring and assessments for progression, if the product is well tolerated and the subject has stable disease or better.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, age ≥ 18 years and ≤75, at the time of study entry.
2. Histologically or cytologically documented advanced colorectal carcinoma with unresectable liver metastasis (existence of extrahepatic metastasis is acceptable).
3. Previously received 2 lines of standard chemotherapy, including 5-FU, oxaliplatin, and irinotecan.
4. Subjects must have at least one measurable lesion per RECIST v1.1.
5. Eastern Cooperative Oncology Group (ECOG) Performance Score of 0 or 1.
6. Estimated life expectancy of ≥12 weeks.
7. Adequate organ functions verified by laboratory tests within 7 days before the first intervention, including bone marrow, liver and kidney function, and coagulation function
8. Female subjects of childbearing potential who are sexually active with a nonsterilized male partner must use an acceptable method of contraception from screening, and must agree to continue using such precautions for 90 days after the final dose of investigational product.
9. Written and signed informed consent.

Exclusion Criteria:

1. ANC<1.5×10*9/L, PLT<80×10*9/L, or Hb<9g/dL; no blood infusion within 2 weeks.
2. TBil>2.5 × ULN.
3. AST or ALT>5 × ULN.
4. Serum Cr>1.5 × ULN, or CrCl<50 ml/min (calculated by Cockcroft-Gault equation)
5. APTT or PT> 1.5 × ULN.
6. Clinically significant electrolyte abnormalities determined by investigators.
7. Proteinuria ≥ 2+ (1.0g/24hr).
8. Hypertension that cannot be controlled by drugs, which is specified as: systolic blood pressure ≥ 140 mmHg and / or diastolic blood pressure ≥ 90 mmHg
9. Active gastrointestinal ulceration, ulcerative colitis, or gastrointestinal bleeding; potential gastrointestinal bleeding or perforation determined by investigators.
10. History of arterial thrombosis or deep venous thrombosis within 6 months before enrollment; evidence of hemorrhagic tendency or receiving anticoagulant therapy within 2 months before enrollment.
11. Stroke or transient cerebral ischemia occurred within 12 months before enrollment.
12. History of cardiovascular disease within 6 months before enrollment, including congestive heart failure (NYHA grade>2), acute myocardial ischemia, severe/unstable angina or CABG; or LVEF<50%.
13. Uncontrollable malignant ascites, pleural effusion, or pericardial effusion (determined by investigators).
14. Previous treated with VEGFR inhibitors.
15. Other malignant tumors in the past 5 years, except skin basal cell or squamous cell carcinoma after radical surgery, or cervical carcinoma in situ.
16. Evidence of CNS metastasis.
17. Active infection, such as acute pneumonia, active stage of HBV/HCV.
18. Pregnant or lactating women.
19. By judgment of the investigator, there are concomitant diseases that seriously endanger the safety of the patient or affect the completion of the study.
20. Severe mental illness.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Estimated)
Dates: Start 2022-02-25 (Actual); Primary Completion 2023-07-31 (Estimated); Study Completion 2024-10-31 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival (PFS) | Up to 2 years
  Progression-free survival is defined as the time from the start of treatment HAIC until the first documentation of disease progression or death due to any cause, whichever occurs first.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | Up to 2 years
  The ORR is defined as the proportion of subjects with confirmed CR or confirmed PR, based on RECIST Version 1.1.
Duration of Response (DoR) | Up to 2 years
  Duration of response is defined as the duration from the first documentation of objective response to the first documented disease progression or death due to any cause, whichever occurs first.
Overall Survival (OS) | Up to 2 years
  Overall survival is defined as the time from the start of treatment with HAIC until death due to any cause.

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Cancer Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No